CLINICAL TRIAL: NCT07031856
Title: Comparison of Clinical Performance of Partial Restorations Fabricated With Three-Dimensional Printer and CAD-CAM: A Split-Mouth Randomized Clinical Trial
Brief Title: Comparison of Clinical Performance of Partial Restorations Fabricated With Three-Dimensional Printer and CAD-CAM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Yaren Cosgun, Research Assistant, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: T.C. Ç.Ü BAP
Record Dates: First submitted 2025-05-20; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Dental Caries; Dental Restoration, Permanent; Tooth Diseases
MeSH Terms: conditions — Dental Caries; Tooth Diseases | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D printer partial crown (Experimental): Participant with restoration produced with 3D printer
  Interventions: Other: 3D printer partial crown
- Cad-Cam partial crown (Other): Participant with restoration produced with Cad-Cam
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: 3D printer partial crown — Comprasion of partial restorations made with 3D printer
  Arms: 3D printer partial crown
Other: Treatment as usual — Cad-cam printer partial crown
  Arms: Cad-Cam partial crown

SUMMARY:
The aim of this clinical study is to compare CAD-CAM and 3D restorations in individuals with two hard tissue losses or restorations in their mouths. The main question it aims to answer is: Is there a difference between CAD-CAM and 3D restorations according to FDI criteria? Researchers will compare participants to see if there is a difference between the two restorations according to FDI criteria. In this split-mouth study, participants will be randomized to receive a CAD-CAM partial restoration on one tooth and a 3D partial restoration on the other tooth.

ELIGIBILITY:
İncluiding:

-- Patients with periodontally stable and appropriate oral hygiene habits without serious systemic diseases that preclude restoration. - Male and female patients with hard tissue loss in their mouth or with 2 teeth in need of restoration replacement (eligibility for split-mouth design). - People who can comply with the treatment and volunteer for follow-up for 2 years-

Exclusion Criteria:

Patients with systemic conditions that may affect the study process (e.g. diabetes, autoimmune diseases).

* Patients with excessive bruxism or parafunctional habits.
* Pregnant or lactating women.
* Patients with gum disease or severe bone loss.
* Patients with a history of allergic reactions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Clinical performance of dental restorations evaluated using FDI World Dental Federation criteria | Baseline, six months, 12 months
  Esthetic Properties Color match (shade stability) Surface staining Translucency/opacity Anatomical form preservation Functional Properties Fracture and retention Marginal adaptation (gap formation) Wear resistance Occlusal contact stability Biological Properties (Newly added) Postoperative hypersensitivity (pulp reactions) Secondary caries development Periodontal response (gingival inflammation, bleeding on probing) Tooth integrity (adjacent tooth structure)

IPD SHARING:
Plan to Share IPD: Yes